CLINICAL TRIAL: NCT06758986
Title: Patients With Subacromial Shoulder Pain and Gender
Brief Title: Is Gender a Factor in Patients With Subacromial Shoulder Pain?
Status: Enrolling by invitation | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Lecturer Dr., Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-010
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Subacromial Pain Syndrome
Keywords: Subacromial Shoulder Pain; functionality; disability; position sense

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group

SUMMARY:
This study aimed to investigate the effects of gender on pain, functionality, range of motion, disability level and position sense parameters in patients with subacromial shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-65
2. Being diagnosed with unilateral subacromial impingement syndrome
3. Not having received steroid injections or physical therapy for shoulder problems in the last 6 months
4. Having painful shoulder pain for the last 3 months
5. Being willing to participate in the study

Exclusion Criteria:

1. Having a rheumatic, neurological, cardiovascular, psychiatric or systemic disorder
2. Having a surgical operation on the shoulder, cervical and thoracic region
3. Having a neurological deficit, fracture or history of fracture in the upper extremity
4. Having cervical radiculopathy
5. Having communication problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted with patients who apply to Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center with complaints of shoulder pain and who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-08-22 (Estimated); Study Completion 2025-09-17 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 20 weeks

SECONDARY OUTCOMES:
Quick DASH | 20 weeks
SPADI | 20 weeks
The laser-pointer assisted angle reproduction test | 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No